CLINICAL TRIAL: NCT02378636
Title: Clinical Investigation of the Modified Rayner Monofocal Aspheric 600C (With Axis Marks) Intraocular Lens
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never initiated
Sponsor: Rayner Intraocular Lenses Limited (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 600C-EU-401; CFLX-2501 (Other: CRO Reference)
Record Dates: First submitted 2015-02-19; First posted 2015-03-04 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2015-11

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 600S (Experimental): Modified 600C (axis marks) monofocal aspheric intraocular lens
  Interventions: Device: 600S

INTERVENTIONS:
Device: 600S — Monofocal Aspheric Intraocular Lens (IOL)
  Other Names: Modified 600C (axis marks)

SUMMARY:
This will be a prospective, open-label, 125 subject (maximum), two-year multicentre investigation to assess the safety, effectiveness and rotational stability of the modified 600C (axis marks) intraocular lens (IOL) in subjects undergoing cataract extraction.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥21 years of age.
* Cataract for which phacoemulsification extraction and posterior IOL implantation has been planned for the operative eye.
* Best corrected distance visual acuity (BCDVA) projected to be better than 20/30 (+0.18 logMAR) in the operative eye after cataract removal and IOL implantation.
* Calculated IOL power requirement within the range +8.0 to +34.0D
* If present, subject must have corneal astigmatism of <1.50 D in the operative eye.
* Expected dilated pupil size ≥ 5.0 mm in diameter to visualise the axis markings
* Subject must provide written informed consent.
* Subject must be able to return for scheduled follow-up examinations for 24 months after surgery.

Exclusion Criteria:

* History of ocular trauma or prior ocular surgery in the operative eye.
* Microphthalmia
* Corneal decompensation or endothelial insufficiency
* Pseudo exfoliation
* Pars planitis
* Subjects with diagnosed degenerative visual disorders in the operative eye (e.g.,macular degeneration or other retinal disorders) that are predicted to cause future visual acuity losses to a level of 20/30 (+0.18 logMAR) or worse.
* Inability to achieve secure placement in the designated location e.g. absence of a secure peripheral anterior capsule, zonule laxity or dehiscence; posterior synechiae to the capsular bag
* Active ocular disease in the operative eye, e.g., clinically significant dystrophy, chronic severe uveitis, proliferative diabetic retinopathy, or chronic glaucoma.
* Concurrent participation in another drug or device investigation.
* Patients who are expected to require retinal laser treatment.
* Females who are pregnant, nursing or plan to become pregnant during the study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Distance Visual Acuity (BCDVA) | 180 Day
  Best Corrected Distance Visual Acuity
Rotational Stability | 180 Day
  IOL rotation will be measured through retro-illumination photography between 0-3 hours post-operatively and this will be compared with images from Day 120-180 to determine degree of IOL rotation in accordance with ISO-11979-7:2014 requirements

CONTACTS AND LOCATIONS:
Overall Officials: Mark Packer, MD, Study Chair — Consultant
Locations (1):
- Contact Rayner Intraocular Lenses Limited for Locations, Hove, East Sussex, United Kingdom